CLINICAL TRIAL: NCT06034600
Title: Effect of Augmented Low-dye Taping and Exercise on Plantar Pressure, Navicular Drop and Foot Posture in Pes Planus
Brief Title: Effect of Augmented Low-dye* Taping and Exercise on Plantar Pressure, Navicular Drop and Foot Posture in Pes Planus
Acronym: Ald
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Asli Oren, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/4027; 0000-0002-5941-1619 (Other: Orcid)
Record Dates: First submitted 2023-03-21; First posted 2023-09-13 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Pes Planus
Keywords: exercise; flat foot; Augmented Low-dye; navicular drop; plantar pressure
MeSH Terms: conditions — Flatfoot; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Experimental, single-blind randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise and taping (Experimental): Individuals in this group are planned to practice exercise together with taping therapy for eight weeks.
  Interventions: Other: taping; Other: exercise
- exercise (Experimental): Individuals in this group are planned to receive only exercise practice for eight weeks.
  Interventions: Other: exercise

INTERVENTIONS:
Other: taping — Taping will be applied to the exercise and taping group after the exercises with theraband. Other exercises that are not performed will be performed with the tape on the skin.The application will be repeated three days a week for eight weeks.
  Arms: exercise and taping
Other: exercise — Stretching and strengthening exercises will be applied to both groups three days a week for 8 weeks.The exercises performed with theraband will be performed in the same way in both groups. While the other exercises will be done after taping in the "taping and exercise group", the "exercise group" will be done without taping.

SUMMARY:
Introduction: Pes planus is a deformity that affects the foot-ankle muscle complex as well as passive components of the foot such as bones and ligaments. Various approaches such as taping methods and exercise training are being investigated in the treatment of pes planus. The effect of the applied methods and their superiority over each other are still unclear. The effect of banding methods varies according to the band type and technique. Exercise methods currently focus on the intrinsic and extrinsic muscles of the foot. Pedobarographic evaluations are also performed in addition to clinical evaluations to evaluate the effectiveness of treatments.

Objective: It is planned to compare the effects of reinforced low-dye taping method, which is one of the rigid taping techniques used in the treatment of pes planus, and exercise training on foot plantar pressure, navicular drop and foot posture.

Material and method: 34 individuals with pes planus between the ages of 18-25 will be included in the study, which was designed as a single-blind randomized study. The universe of our study will be Lokman Hekim University Faculty of Health Sciences and Institute of Health Sciences. The whole universe will be tried to be reached and individuals who meet the inclusion criteria will be selected from the relevant universe. Consent form will be obtained from individuals who are deemed eligible to participate in the study. Pes planus evaluation; It will be done using the navicular drop test and the foot posture index. In order for the physical activity levels of the groups to be homogeneous, after stratified sampling, individuals will be randomly assigned to the exercise groups by taping and exercise with the closed envelope method. Evaluations will be made to each group at the beginning, at the eighth and twelfth week. Static evaluation of the foot will be made using navicular drop and foot posture index, and pedobarographic analysis will be done using a foot analyzer.

Conclusion: The effects of taping and exercise training on foot static and plantar pressure measurements will be interpreted.

DETAILED DESCRIPTION:
For taping application, intermittent taping will be done by the same researcher on the foot with pes planus three times a week. The applied hard taping technique will be applied continuously for eight weeks. The group that will perform exercises together with the taping treatment will perform the exercises with the resistance band without taping and then do the other exercises after the taping application. The applied taping will remain on the skin as long as it can until the next taping day. Individuals will be asked to note the length of stay of the tape on the skin. The exercises will be done three days a week for eight weeks. After verbal information about the research protocol to be applied, practical training will be given for the exercises. In the banding application, reinforced low-dye (ALD) technique, one of the hard banding techniques, will be applied. A hard tape will be used on the individuals by the same researcher throughout the study. With the tape application, to the participants; Information will be given about physical activity, shoes and issues that should be considered in daily life.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-25
* Navicular drop (ND) test >10 mm
* Foot posture index ≥6
* Individuals in the 1st and 2nd category according to the international physical activity survey
* Individuals who volunteered to participate in the study

Exclusion Criteria:

* Presence of systemic, neurological, rheumatological or orthopedic problems that may affect the lower extremity
* Individuals who are allergic to the tape to be used
* Individuals who cannot adapt to exercise or taping practices
* Individuals who have received treatment for pes planus in the last 6 months
* Individuals with a BMI ≥ 30
* Presence of pregnancy
* Cases not wanting to take part in the study

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
foot plantar pressure | baseline, at 8 and 12 weeks
  A foot analyzer will be used in the pedobarographic evaluation of the foot.

SECONDARY OUTCOMES:
navicular drop | baseline, at 8 and 12 weeks
  The distance measurement from the ground with the navicular will be measured using the caliper. Three measurements will be taken and the average recorded.
foot posture index | baseline, at 8 and 12 weeks
  Each criterion is scored on a scale ranging from -2 to +2, when the score is between 0 and 5, the foot will be considered neutral and between 6 and +12 as pronation.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Talu, PhD, Study Director — Inonu University
Locations (1):
- Inonu Univercity, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tang M, Wang L, You Y, Li J, Hu X. Effects of taping techniques on arch deformation in adults with pes planus: A meta-analysis. PLoS One. 2021 Jul 2;16(7):e0253567. doi: 10.1371/journal.pone.0253567. eCollection 2021. PMID 34214104
- [Result] Hoang NT, Chen S, Chou LW. The Impact of Foot Orthoses and Exercises on Pain and Navicular Drop for Adult Flatfoot: A Network Meta-Analysis. Int J Environ Res Public Health. 2021 Jul 29;18(15):8063. doi: 10.3390/ijerph18158063. PMID 34360354